CLINICAL TRIAL: NCT00821457
Title: A Within Patient, Placebo Controlled, Proof of Concept Trial to Assess the Efficacy of Juvista in Improving the Appearance of Existing Scars That Are 2-6 Months Old
Brief Title: Juvista in the Non-surgical Improvement of Existing Scars
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Dr James Bush, Renovo
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RN1001-0098
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Scars
Keywords: existing scars the are two to six months old
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): 250ng Juvista vs placebo
  Interventions: Drug: Juvista; Drug: Placebo
- Group 2 (Active Comparator): 500 ng Juvista vs placebo
  Interventions: Drug: Placebo; Drug: Juvista

INTERVENTIONS:
Drug: Juvista — 250ng
  Other Names: Avotermin; Recombinant Transforming Growth Factor Beta 3
  Arms: Group 1
Drug: Placebo — Powder for solution for injection
Drug: Juvista — 500ng
  Other Names: Avotermin; Recombinant Transforming Growth Factor Beta 3
  Arms: Group 2

SUMMARY:
Renovo, a Biopharmaceutical company involved in the development of drugs to improve the appearance of scars and enhance wound healing, are proposing to carry out research in improving the appearance of existing scars that are 2-6 months old using Juvista. Juvista has not previously been administered to pre-existing scars without surgical revision, but it is thought that some beneficial effects seen with Juvista in previous trials may also be seen when administered to existing scars whilst the scar is maturing. This proof of concept study will therefore investigate the effect of Juvista in Caucasian male and female patients when administered to scars that are between two and six months old.

Scarring in the skin can vary hugely between individuals; therefore the most reliable way to assess the efficacy of an improvement of scar appearance is to use a model where each patient acts as their own control. A placebo will also be used for this trial as there are currently no approved pharmaceuticals for the improvement of scarring.

A total of 20 patients will be allocated to one of two dosing groups. Patients who enter the study will have linear scars resulting from broken skin (e.g. trauma, surgery) between 7 and 20cm in length, as well as meeting other specific criteria. The scar to be treated will be divided into two equal segments. Each segment will receive an intradermal injection of Juvista or placebo on Day 0 and 24 hours later.

The measure of change in scar appearance will be performed using colour analysis which will assess the change in colour between the Juvista treated segments versus the placebo treated segment of the scar, with reference to the surrounding skin within each patient.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Caucasian patients aged 18-45 years who have provided written informed consent.
* A body mass index between 15 and 35 kg/m2 (calculated using Quetelet's index [weight (kg)/height m2]
* Patients with, in the opinion of the Investigator, clinically acceptable results for the laboratory tests specified in the trial protocol (see Section 6.4.2). All laboratory tests must be performed within 28 days of the first trial dose administration.
* Female patients of child bearing potential who are using a highly effective method(s) of contraception and agree to do so from at least the screening visit until one month after administration of the final study dose. For the purposes of the protocol, highly effective method(s) of contraception will be defined as consistently and correctly used implants, injectables, combined oral contraceptives, sexual abstinence or a vasectomised partner
* The scar to be treated is 2-6 months old at Day 0.
* The scar is linear.
* The scar to be treated is symmetrical in appearance around the mid-line.
* The scar to be treated is between 7cm and 20cm in length and a maximum of 1cm in width.
* The scar to be treated runs along a flat surface which is in the same focal plane and suitable for accurate medical photography.

Exclusion Criteria:

* Patients who on direct questioning and / or physical examination, have evidence of any past or present clinically significant medical condition that would impair wound healing including :

  * Significant rheumatoid arthritis.
  * Significant hepatic impairment (LFTs >3 times upper limit of normal).
  * Inadequately or uncontrolled congestive heart failure.
  * Currently active malignancy or history of any malignancy in the 5 years prior to the screening visit.
  * Immunosuppression or chemotherapy in the twelve months prior to the screening visit.
  * A history of radiotherapy to the study scar area.
  * Diabetes mellitus (unless controlled by diet and exercise alone).
  * A bleeding disorder or current use of anti-thrombotic therapy (aspirin, ticlopidine and clopidogrel are permitted).
* Patients with a creatinine clearance (CLcr) of 80ml/min or less. Creatinine clearance will be determined from the serum creatinine level at pre-study screening using the following formula :

  o CLcr = (140-age (years)) x weight(kg)/ 72 x serum creatinine (mg/dL) { x 0.85 for females }
* Patients with a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* Patients with a history of clinically relevant allergy, hypersensitivity, angioedema, or anaphylaxis.
* Patients with a progressive neurological condition including Parkinson's disease, Alzheimer's disease and uncontrolled epilepsy.
* Patients with a known history of chronic viral infection (Hepatitis, HIV) or ongoing active infection.
* Patients with bleeding disorders including haemophilia, purpura or thrombocytopenia or receiving anticoagulants (e.g. warfarin, coumadin).
* Patients with an ongoing psychiatric condition requiring treatment or psychosis (including depression with psychosis, bipolar disease and schizophrenia.
* Patients with a history of clinically significant hypersensitivity to any of the drugs, surgical markers or surgical dressings to be used in this trial.
* Patients who are taking, or have taken, any investigational drugs within 3 months prior to the screening visit.
* Patients undergoing investigations or changes in management for an existing medical condition.
* Female patients who are breast feeding, or intending to become pregnant or breast feed during the study period (subjects must be using adequate contraception and have a negative pregnancy test at screening).
* Female patients who have had any change in their oral contraceptive medication (if applicable) in the 2 months prior to screening, or anticipate any change during study participation
* In the opinion of the Investigator, a patient who is not likely to complete the trial for whatever reason.
* Patients with a history of substance abuse or dependency (a history of recreational use of cannabis is acceptable assuming a negative urine test for cannabis at screen. Patients who have had a history of alcohol abuse but have been dependency free for 12 months will still be eligible).
* Patients who on direct questioning and physical examination have a history or evidence of keloid scarring.
* Patients with additional scars less than 3cm away from the scar to be treated.
* The scar to be treated is a facial scar.
* Patients who are involved in ongoing litigation in connection with the scar to be treated.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy variable is the change in scar appearance at 6 months post treatment, assessed by calculating the colour difference between the treated scar sections with reference to the surrounding skin. | 6 months post treatment

SECONDARY OUTCOMES:
The secondary efficacy variable is the difference in scar appearance between active and placebo treated segments at 6 months post treatment as assessed using a global scar comparison scale | 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: James Dr Bush, MBChB MRCS, Principal Investigator — Renovo
Locations (1):
- Renovo Clinical Trial Unit, Manchester, Greater Manchester, United Kingdom